CLINICAL TRIAL: NCT03201393
Title: A Single Site, Phase 2B, Randomized, Double-Blind, Study to Assess the Efficacy, Safety, and Tolerability of Low-Dose Naltrexone and Acetaminophen Combination vs. Placebo in the Treatment of Chronic Low Back Pain (ANODYNE-4)
Brief Title: Low-Dose Naltrexone and Acetaminophen Combination in the Treatment of Chronic Low Back Pain (ANODYNE-4)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Allodynic Therapeutics, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ANODYNE-4
Record Dates: First submitted 2017-06-16; First posted 2017-06-28 (Actual); Last update posted 2021-04-14 (Actual); Status verified 2018-04

CONDITIONS: Chronic Low Back Pain; Lumbar Radiculopathy
Keywords: Back pain; Neuropathic Pain; Radiculopathy; Allodynia
MeSH Terms: conditions — Radiculopathy; Back Pain; Neuralgia; Hyperalgesia | interventions — Naltrexone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Low-Dose Naltrexone and Acetaminophen Combination (Experimental)
  Interventions: Drug: Low-dose naltrexone and acetaminophen combination
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Low-dose naltrexone and acetaminophen combination — Twice a day
  Arms: Low-Dose Naltrexone and Acetaminophen Combination
Drug: Placebo — Twice a day
  Arms: Placebo

SUMMARY:
Treatment of chronic low-back pain with low-dose naltrexone and acetaminophen combination: a small, randomized, double-Blind, and placebo-controlled clinical trial with an open-label extension for none-responders

ELIGIBILITY:
Inclusion Criteria:

1. The patient is a male or female 18 years of age or older.
2. A clinical diagnosis of nonmalignant, chronic low back pain (CLBP). LBP, as defined by Quebec Task Force in class 1 - pain without radiation and class 2 - pain with proximal radiation above the knee. CLBP is defined as being present for at least several hours a day, at least half the days in the previous 6 months, and being the principal pain condition. (In accordance with the NIH 2013 Task Force on Research Standards for Chronic Low Back Pain).
3. The 24-hour average pain intensity (API) mean score for the baseline period is ≥ 4 and ≤ 8, [measured on the 11-point (0-10) numeric rating scale (NRS)] with each individual score ≥ 3. In addition, the Oswestry Disability Index (ODI) score during the Randomization Visit is ≥ 30% and ≤ 60%.

5. The patient agrees to refrain from taking opiate medications from Visit 1 to 7 days after the last dose of the study drug.

6. The patient agrees to limit their rescue pain medications to acetaminophen 2000 mg per day for the duration of the study.

7. The patient is willing and able to discontinue use of non-pharmacological pain management modalities (e.g. TENS, physical therapy, chiropractic manipulations, biofeedback, and acupuncture) for the duration of the study.

8. The patient has been taking a stable dose of a medication with pain prevention potential for at least 6 weeks prior to the screening visit and agrees to not start, stop, or change the dose of any medication with pain prevention potential during the study period. (E.g., tricyclic antidepressants, anticonvulsants, selective serotonin reuptake inhibitors (SSRIs), serotonin-norepinephrine reuptake inhibitors (SNRIs), herbal preparations (e.g. feverfew or St. John's wort)). Botulinum toxin injections and steroid injections to the spine must be discontinued six months prior to Visit 1.

9. The patient is able to complete study questionnaires, comply with the study requirements and restrictions, and willing to provide written informed consent and authorize HIPAA.

10. The patient agrees not to undergo any elective surgery, including spine surgery or injections to the spine (e.g. botulinum toxin, steroid, etc.) for the duration of the study.

11. The Female patient who is premenopausal or postmenopausal less than 1 year, or have not had surgical sterilization (i.e., tubal ligation, partial or complete hysterectomy) must have a negative serum pregnancy test, be non-lactating, and commit to using adequate and reliable contraception throughout the study (e.g., barrier with additional spermicidal, intra-uterine device, hormonal contraception). Male patients must be surgically sterile or commit to the use of 2 different methods of birth control during the study and for 28 days after the study.

Exclusion Criteria:

1. The patient has any condition consistent with Quebec Task Force Classification 3-11.
2. The patient has another painful condition that may require analgesic medications, occurring regularly or intermittently (e.g. menstrual pain, carpal tunnel syndrome, arthritis, tendinitis, etc.).

The patient has concomitant migraine unless he/she treats migraine attacks only with ergotamine or triptans.

4. Regular use of the following medications for any reason: acetaminophen, non-steroidal anti-inflammatory drugs (NSAIDs), antipsychotic drugs, monoamine oxidase inhibitors, muscle relaxants, blood thinning medications (e.g., warfarin or heparin), or cannabinoids. Low-dose aspirin for cardiovascular disease prophylaxis is permitted.

5. Diagnosis of any concurrent medical or psychiatric condition; this includes, chronic unstable debilitating diseases such as Parkinson's disease, multiple sclerosis, cancer, significant renal impairment, significant hepatic impairment, etc.

6. The patient has a history or diagnosis of moderate-to-severe hepatic or renal impairment (>2 × the upper limit of normal [ULN] for alanine transaminase or aspartate transaminase. ≥1.5 × ULN for Alkaline Phosphatase, bilirubin, BUN, or Creatinine). (Patients with elevated bilirubin level due to Gilbert's syndrome are allowed).

7. The patient has a history of the previous 5 years of abuse of any drug, prescription, illicit, or alcohol.

8. The Female patient is pregnant or breastfeeding. The Male patient is not practicing 2 different methods of birth control with their partner during the study, and for 28 days after the investigational drug last dose or will not remain abstinent during the study, and for 28 days after the last dose.

9. The patient has known-hypersensitivity to components of the investigational drug.

10. Participation in another study with an investigational drug within 30 days before Visit 1 or during the study.

11. The patient is in the opinion of the investigator, unsuitable to participate in this study for any other reason.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2017-08-15 (Actual); Primary Completion 2018-07-26 (Actual); Study Completion 2018-07-26 (Actual)

PRIMARY OUTCOMES:
The change from baseline in mean 7-day, 24-hour Worst Pain Intensity (WPI). | From baseline to the last 7 days of the 12-week double-blind treatment period.
  The mean weekly WPI score will be derived from assessments recorded by patients daily at bedtime. The WPI score is measured on the 11-point (0-10) Numeric Rating Scale (NRS), (0=no pain, 10=worst possible pain).

SECONDARY OUTCOMES:
The change from baseline in mean 7-day, 24-hour Average Pain Intensity (API). | From baseline to the last 7 days of the 12-week double-blind treatment period.
  The mean weekly API score will be derived from assessments recorded by patients daily at bedtime. The API score is measured on the 11-point (0-10) NRS.
Proportion of patients with 50% or more reduction in 7-day, 24-hour Worst Pain Intensity (WPI). | From baseline to the last 7 days of the 12-week double-blind treatment period.
  The mean weekly WPI score will be derived from assessments recorded by patients daily at bedtime. The WPI score is measured on the 11-point (0-10) NRS.
The change from baseline in mean 7-day, 24-hour Right Now Pain Intensity (NPI). | From baseline to the last 7 days of the 12-week double-blind treatment period.
  The mean weekly NPI score will be derived from assessments recorded by patients daily at bedtime. The NPI score is measured on the 11-point (0-10) NRS.
The change from baseline in mean 7-day, 24-hour Pain-Related Interference (PRI) with day-to-day activities. | From baseline to the last 7 days of the 12-week double-blind treatment period.
  The mean weekly PRI score will be derived from assessments recorded by patients daily at bedtime. The PRI score is measured on the 11-point (0-10) NRS.
The change from baseline in mean 7-day, 24-hour pain-related sleep interference (PRSI). | From baseline to the last 7 days of the 12-week double-blind treatment period.
  The mean weekly PRSI score will be derived from assessments recorded by patients daily at bedtime. The PRSI score is measured on the 11-point (0-10) NRS.
Change from baseline in the mean number of rescue medications used. | From baseline to the last 7 days of the 12-week treatment period.
  Rescue medications use will be derived from daily recordings by patients.
Change from baseline in the mean Oswestry Disability Index (ODI). | From baseline to the last 7 days of the 12-week double-blind treatment period.
  Patients will complete the ODI instrument during site visits (%).
Change from baseline in the mean Pittsburgh Insomnia Rating Scale-20 (PIRS-20). | From baseline to the last 7 days of a 12-week double-blind treatment period.
  Patients will complete the PIRS-20 instrument during site visits (0-60).

OTHER OUTCOMES:
Comparison of the proportion of patients who experienced adverse events. | Completion of the treatment period at 12 weeks.
  Defined as any untoward medical occurrences, regardless of their suspected cause.

CONTACTS AND LOCATIONS:
Overall Officials: Annette Toledano, M.D., Principal Investigator — Allodynic Therapeutics, Inc
Locations (1):
- Annette C. Toledano, M.D., North Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No